CLINICAL TRIAL: NCT01926249
Title: A Cohort of Outpatients From French Research Memory Centers in Order to Improve Knowledge on Alzheimer's Disease and Related Disorders
Acronym: MEMENTO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Fondation Plan Alzheimer (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/47
Record Dates: First submitted 2013-08-16; First posted 2013-08-20 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer's Disease (AD) and Related Disorders
Keywords: Alzheimer's disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood sampling
  * Lumbar puncture (samples without DNA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals at high risk of developing Alzheimer's dementia: * 2000 participants with a newly identified cognitive deficit defined as performing worse than one standard deviation to the mean in one or more cognitive domain (memory, language, praxis, visuospatial abilities, attention and executive functions), not demented.
  * 300 participants with an isolated cognitive complaint and an age of 60 years or more.

SUMMARY:
A Multicenter national prospective cohort study including at least 2300 individuals consecutively recruited from French Research Memory Centers and followed-up over 5 years.

DETAILED DESCRIPTION:
The increasing incidence of Alzheimer's disease (AD) and related disorders with the change in the world age demographic is a source of major public health concern. Early and accurate identification of individuals at high risk of Alzheimer's Disease has become a priority. Over the last years, research has focused on the concept of "Mild Cognitive Impairment" which happens to be a heterogeneous condition as, depending on the studies, Mild Cognitive Impairment patients' conversion rates to dementia range from 2 to 15 percent per year. A study of the full range of stages of evolution, from preclinical stage, to clinical expression of dementia or death is therefore of utmost importance to improve our knowledge on AD and trigger the development of new treatments, especially if between stages transition can be related to neuroimaging (either structural or molecular), biological (Cerebro-Spinal Fluid, serum or plasma) or vascular damages markers. However, if all the above markers have been shown to be individually associated with worsening of cognitive status, no prior study has simultaneously explored the association of a large panel of risk factors and biomarkers with the progression through early signs of cognitive impairment until AD in a large sample of study participants. In parallel to improving the knowledge on AD, it is also important to better estimate the social and economic burden of AD and their consequences on the individuals and their circle and how they evolve from early phase (pre-clinical) of the disease to the most severe stages.

This cohort, solution to the item 29 of the Plan Alzheimer 2008-2012, has been developed according to the initial memorandum of understanding prepared by the "Comité Plan Cohortes" of the Fondation Plan Alzheimer, and taking on board comments provided by the Scientific Advisory Board (July 2010) of the Fondation Plan Alzheimer and the whole working groups constituted for the preparation of the pilot phase: clinicians, neuro-imaging specialists, biologists, social sciences researchers (from June 2010). The cohort is built to fulfil the guiding principles as follows:

* It should be scientifically original and identify hypothesis-driven research, allowing a corpus of new or confirmatory knowledge of a high-level of evidence to be acquired. In addition, the infrastructure (standardised collection of socio-demographic, clinical, imaging, biological data) may allow to respond, in a timely manner, to additional questions that may emerge over time;
* An interdisciplinary approach is set up as the condition of individuals affected by neurodegenerative dementias involves clinical and biological aspects but also environmental, social and economic components;
* While pursuing its own original scientific objectives, the cohort should have the potential for a comparison with other equivalent cohorts around the world.

This cohort will be including individuals at high risk of developing a neurodegenerative dementia. As such, the cohort is aiming at providing results with an expected impact for those individuals of the same profile, as well as their caregivers and their case management.

One expected impact is to increase knowledge on the progression from early signs of cognitive impairment to AD and estimate associations between these signs and level of biomarkers assessed through imaging or blood or CSF samples. Another major expected impact is to standardise and harmonise protocols in terms of clinical and neuro-psychological examinations, biological markers, neuroimaging markers, diagnosis of dementia, support to caregivers and informants.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Having at least a light cognitive deficit defined as performing worse than one standard deviation to the mean (compared to age and educational norms) in one or more cognitive domains (assessed from a neuropsychological tests battery exploring memory, language, praxis, vision, executive functions); this deviation being identified for the first time by tests performed less than 6 months preceding date of inclusion
* Or having isolated cognitive complaint regardless of its duration while being 60 years and older
* Clinical Dementia Rating scale <=0.5 and not demented
* Visual and auditory acuity adequate for neuropsychological testing
* Having signed an informed consent
* Being affiliated to health insurance

Exclusion Criteria:

* Being under guardianship
* Residence in skilled nursing facility
* Pregnant or breast feeding women
* Alzheimer's disease caused by gene mutations
* Meeting brain MRI exclusion criteria (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body) or refusing MRI
* Having a neurological disease such as: treated epilepsy, treated Parkinson's disease, Huntington disease, brain tumour, subdural haematoma, progressive supranuclear palsy, history of head trauma followed by persistent neurological deficits
* Stroke that has occurred in the last three months
* Schizophrenia history (DSM-IV criteria)
* Illiteracy, is unable to count or to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from French Research Memory Centers with at least a light cognitive deficit defined as performing worse than one standard deviation to the mean in one or more cognitive domains or an isolated cognitive complaint regardless of its duration while being 60 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 2325 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Progression to clinical dementia stage according to standardized classifications (DSM-IV for dementia and NINCDS-ADRDA for Alzheimer's disease) | Each 6 months from baseline for 5 years (M60)

SECONDARY OUTCOMES:
Mortality | Each 6 months from baseline for 5 years (M60)
Loss of autonomy based on functional activity assessment | Each 6 months from baseline for 5 years (M60)
Institutionalisation | Each 6 months from baseline for 5 years (M60)
Speed of cognitive decline based on change in cognitive performances | Each 6 months from baseline for 5 years (M60)
Cardiovascular event (Stroke and Coronary events) | Each 6 months from baseline for 5 years (M60)
Quality of life | Each 6 months from baseline for 5 years (M60)
Prodromal AD (Pre-symptomatic dementia) | Each 6 months from baseline for 5 years (M60)
Longitudinal evolution of biomarkers measured from blood, Cerebro-Spinal Fluid (CSF), structural neuroimaging (MRI) and molecular neuroimaging (18F-FDG PET) | Each 6 months from baseline for 5 years (M60)

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve CHENE, Prof, Principal Investigator — CIC-EC7 - ISPED - CHU de Bodeaux; Geneviève CHENE, Prof, Study Chair — CIC-EC7 - ISPED - CHU de Bordeaux; Carole DUFOUIL, Director, Study Director — CIC-EC7 - ISPED - CHU de Bordeaux
Locations (29):
- France (29):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU de Besançon, Besançon
  - AP-HP - Avicenne, Bobigny
  - CHU de Bordeaux - Pellegrin, Bordeaux
  - CHU de Bordeaux - Hôpital Xavier-Arnozan, Bordeaux
  - CHU de Brest, Brest
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpitaux civils de Colmar, Colmar
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - Hospices civils de Lyon, Lyon
  - AP-HM, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - AP-HP - Hôpital BROCA, Paris
  - AP-HP - Hôpital LARIBOISIERE, Paris
  - Ap-Hp La Pitié-Salpêtrière, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne - Hôpital de la charité, Saint-Etienne
  - CHU de Saint-Etienne - Hôpital Nord, Saint-Etienne
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse - Hôpital Purpan, Toulouse
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Lespinasse J, Dufouil C, Proust-Lima C. Disease progression model anchored around clinical diagnosis in longitudinal cohorts: example of Alzheimer's disease and related dementia. BMC Med Res Methodol. 2023 Sep 5;23(1):199. doi: 10.1186/s12874-023-02009-0. PMID 37670234
- [Derived] Blanc F, Bouteloup V, Paquet C, Chupin M, Pasquier F, Gabelle A, Ceccaldi M, de Sousa PL, Krolak-Salmon P, David R, Fischer C, Dartigues JF, Wallon D, Moreaud O, Sauvee M, Belin C, Harston S, Botzung A, Albasser T, Demuynck C, Namer I, Habert MO, Kremer S, Bousiges O, Verny M, Muller C, Philippi N, Chene G, Cretin B, Mangin JF, Dufouil C. Prodromal characteristics of dementia with Lewy bodies: baseline results of the MEMENTO memory clinics nationwide cohort. Alzheimers Res Ther. 2022 Jul 19;14(1):96. doi: 10.1186/s13195-022-01037-0. PMID 35854388
- [Derived] Dufouil C, Dubois B, Vellas B, Pasquier F, Blanc F, Hugon J, Hanon O, Dartigues JF, Harston S, Gabelle A, Ceccaldi M, Beauchet O, Krolak-Salmon P, David R, Rouaud O, Godefroy O, Belin C, Rouch I, Auguste N, Wallon D, Benetos A, Pariente J, Paccalin M, Moreaud O, Hommet C, Sellal F, Boutoleau-Bretonniere C, Jalenques I, Gentric A, Vandel P, Azouani C, Fillon L, Fischer C, Savarieau H, Operto G, Bertin H, Chupin M, Bouteloup V, Habert MO, Mangin JF, Chene G; MEMENTO cohort Study Group. Cognitive and imaging markers in non-demented subjects attending a memory clinic: study design and baseline findings of the MEMENTO cohort. Alzheimers Res Ther. 2017 Aug 29;9(1):67. doi: 10.1186/s13195-017-0288-0. PMID 28851447